CLINICAL TRIAL: NCT00385294
Title: Role of B2 Adrenergic Receptors in Labor Pain
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela Flood, Professor of Anesthesiology, Columbia University
Other Study IDs: AAAB3535
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Pain; Pain Threshold; Labour Pain
Keywords: Genetic; pain; obstetrical
MeSH Terms: conditions — Pain; Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA identified by subject number will be retained for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to understand why labor is more painful for some women compared to others. The study will study whether a woman's baseline pain sensitivity, beta2 adrenergic receptor genotype is related to her pain in labor for the birth of a first child.

DETAILED DESCRIPTION:
Other than parity, and infant size, the etiology of the great variability in labor pain us unknown. Previous studies have demonstrated that baseline pain sensitivity is related to postoperative pain and narcotic requirement. We hypothesize that baseline pain sensitivity is related to pain in labor. The study will determine baseline sensitivity to heat, cold and pressure as measurement of pain sensitivity. Furthermore, b2 adrenergic genotype has recently been identified as a potential determinant of pain sensitivity. The investigators will determine whether B2 receptor haplotype is an independent predictor of pain experienced in labor.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women
* Third trimester of pregnancy on enrollment

Exclusion Criteria:

* Chronic Pain
* Pain medication utilization
* Large for gestational age baby
* Small for gestational age baby
* Systemic illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nuliparous women anticipating NSVD
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela D. Flood, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Liang DY, Liao G, Wang J, Usuka J, Guo Y, Peltz G, Clark JD. A genetic analysis of opioid-induced hyperalgesia in mice. Anesthesiology. 2006 May;104(5):1054-62. doi: 10.1097/00000542-200605000-00023. PMID 16645459
- [Background] Hsu YW, Somma J, Hung YC, Tsai PS, Yang CH, Chen CC. Predicting postoperative pain by preoperative pressure pain assessment. Anesthesiology. 2005 Sep;103(3):613-8. doi: 10.1097/00000542-200509000-00026. PMID 16129988